CLINICAL TRIAL: NCT02179697
Title: Radiographic and Clinical Outcomes Following Non-operative Versus Operative Treatment of AO Type A3 Fractures: A Prospective, Randomized Clinical Trial With an Observational Component
Brief Title: Randomized Trial With an Observational Component of Non-operative Versus Operative Treatment for AO Type A3 Fractures
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: H Francis Farhadi (Other)
Responsible Party: Sponsor-Investigator, H Francis Farhadi, Assistant Professor, Ohio State University
Organization: Ohio State University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2014H0100
Record Dates: First submitted 2014-06-16; First posted 2014-07-02 (Estimated); Last update posted 2017-01-18 (Estimated); Status verified 2017-01

CONDITIONS: Spinal Fractures
Keywords: Groups:; Group 1 (2 Treatment Arms (Randomized between 2 treatments)); Treatment 1: Surgery + Bracing; Treatment 2: Bracing Alone; Group 2; The patient will decide which group is best for themselves.
MeSH Terms: conditions — Spinal Fractures | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Surgery + Bracing vs. Bracing Alone (Active Comparator): Randomize between 2 treatments:
  Treatment 1: Surgery + Bracing Treatment 2: Bracing alone
  Interventions: Procedure: Surgery + Bracing vs. Bracing Alone
- Patient's choice (Other): Patient will decide which group is best for him/her. The patient will be followed at the same points as Group 1.
  Interventions: Other: Patient's Choice

INTERVENTIONS:
Other: Patient's Choice — Patient chooses between surgery plus bracing or bracing alone. The patient will be followed according to the same schedule as Group 1.
  Arms: Patient's choice
Procedure: Surgery + Bracing vs. Bracing Alone — Surgery + Bracing vs. Bracing Alone
  Arms: Surgery + Bracing vs. Bracing Alone

SUMMARY:
The purpose of this study is to compare surgery plus bracing versus bracing alone. Both groups are considered standard of care treatments. The goal of this study is to determine which group is a better treatment.

DETAILED DESCRIPTION:
Patient must be between 18 and 65 years old and had an acute trauma with an AO type A3 burst fracture (a spinal injury where one of the bony parts of the spine [vertebra] breaks due to immediate and severe compression).

The purpose of this study is to compare surgery plus bracing versus bracing alone. Patients will be followed for 10 years. The investigators will compare patients' x-ray outcomes and clinical outcomes (i.e. how a patient is feeling and how a patient is able to do usual daily activities) as well as patients' immediate and delayed medical and surgical side effects between the 2 study arms. The goal of this study is to determine if treating patients with surgery plus bracing is better than just bracing alone.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-65 years
2. Acute trauma patient with AO Type A3.1-A3.3 fractures of T10-L2
3. Neurologically intact
4. TLICS score of 4
5. Women of childbearing potential must have a negative serum pregnancy test

Exclusion Criteria:

1. Severe poly-trauma (Injury Severity Score >15 and/or intubation required for > 24 hours)
2. Sepsis and/or organ failure
3. Prior instrumented arthrodesis of the thoracolumbar spine
4. Severe co-morbidities (e.g., heart, respiratory, or renal disease)
5. Recent history (<3 years) of concomitant spinal tumor or infection
6. Greater than single level fracture involvement (other than transverse process fractures)
7. AO Type A3 fracture with associated load sharing score ≥7
8. ≥ 30 degrees regional kyphosis on standing
9. History of autoimmune (seronegative) spondyloarthropathy (i.e., ankylosing spondylitis)
10. History of osteoporosis
11. Subjects who are pregnant or plan to become pregnant in the next 24 months. Patients will be advised on the use of contraceptives during this time. Methods include abstinence or two acceptable forms including condoms with spermicide, birth control pills, injections, or an IUD.
12. Co-morbidity requiring medication that may interfere with bone or soft tissue healing (i.e., oral or parenteral glucocorticoids, NSAIDs immunosuppressive agents, methotrexate)
13. Severe morbid obesity (BMI > 40)
14. History of metal sensitivity/foreign body sensitivity
15. History of prior laminectomy at the fracture site
16. Associated scoliotic (> 10°) or pre-existing thoracolumbar kyphotic deformity
17. History of substance abuse (recreational drugs, prescription drugs or alcohol) that could interfere with protocol assessments and/or with the subject's ability to complete the protocol required follow-up
18. Prisoner

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-08; Primary Completion 2017-06 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
Compare radiologic outcomes using regional kyphosis and Evaluate clinical outcomes using questionnaires | 2 years
  Primary Outcome is to compare radiologic and clinical outcomes. These will be measured by regional kyphosis, at 2 years following either non-operative or operative management of thoracolumbar AO type A3.1, A3.2, A3.3 fractures in neurologically-intact patients; and Oswestry Disability Index, at 2 years following either non-operative or operative management of thoracolumbar AO type A3.1, A3.2, A3.3 fractures in neurologically-intact patients.

SECONDARY OUTCOMES:
Compare radiologic outcomes using regional kyphosis | 5 and 10 years
  Secondary outcome is to compare radiologic outcomes, as measured by regional kyphosis, at 5 and 10 years following either non-operative or operative management of thoracolumbar AO type A3.1, A3.2, A3.3 fractures in neurologically-intact patients
Evaluate clinical outcomes using questionnaires | 5 and 10 years
  Secondary outcome is to evaluate clinical outcomes, as measured by the Oswestry Disability Index, at 5 and 10 years following either non-operative or operative management of thoracolumbar AO type A3.1, A3.2, A3.3 fractures in neurologically-intact patients.
Compare global sagittal balance at 3 different time points | 2,5, and 10 years
  Secondary Outcome is to compare global sagittal balance at 2, 5, and 10 years.
Collect data on patient in both groups for 10 years | 10 years
  Secondary Outcome is to record frequency and time to secondary surgical intervention among patients in the bracing group.
Compare Return to work rates over a two year peiord | 3 month, 1 year, and 2 years
  Secondary Outcome is to Compare return-to-work rates at 3 months, 1 year, and 2 years following either non-operative or operative management of thoracolumbar AO type A3.1, A3.2, A3.3 fractures in neurologically-intact patients.
Compare Health Care Cost between both groups over 10 years | 10 years
  Secondary Outcome is to compare health care cost and utilization through extended follow-up period.

CONTACTS AND LOCATIONS:
Overall Officials: Francis Frahadi, MD, PhD, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State Unviersity, Columbus, Ohio, United States